CLINICAL TRIAL: NCT01911611
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study in Healthy Volunteers to Assess the Safety, Tolerability, Pharmacodynamics and the Effect of Food on the Pharmacokinetics of RO6870868
Brief Title: A Study of RO6870868 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NP28628
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- RO6870868 (Experimental)
  Interventions: Drug: RO6870868

INTERVENTIONS:
Drug: RO6870868 — Single ascending doses
  Arms: RO6870868
Drug: placebo — Single ascending doses
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the safety, tolerability, pharmacokinetics of RO6870868 in healthy volunteers. Subjects will be randomized to receive single ascending doses of either RO6870868 or placebo, with or without food.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 65 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Women of non-childbearing potential including women who have undergone hysterectomy or bilateral oophorectomy and postmenopausal females
* Male subjects must be willing to use effective contraception as defined by protocol for the duration of the study and for one month after the last dose of study medication
* Body Mass Index (BMI) at screening of 18 to 32 kg/m2, inclusive
* Non-smokers, or use of < 10 cigarettes (or equivalent nicotine-containing product) per day
* No medical or social conditions that would potentially interfere with the subjects ability to comply with the study visit schedule or the study assessments

Exclusion Criteria:

* Pregnant (positive pregnancy test) or lactating women, and male partners of women who are pregnant or lactating
* History of drug or alcohol abuse within the last year
* History of immunologically mediated disease
* History or symptoms of any significant disease including (but not limited to) neurological, cardiovascular, endocrine, respiratory, gastrointestinal, hepatic, or renal disorder
* Personal or family history of congenital long QT syndrome or sudden death
* Evidence of an active or suspected cancer or a history of malignancy where in the investigator's opinion, there is a risk of recurrence. History of having received any systemic anti-neoplastic (including radiation) or immunomodulatory treatment (including systemic oral or inhaled corticosteroids) </= 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable)
* History of significant psychiatric disease
* Significant acute infection, e.g., influenza, local infection, acute gastrointestinal symptoms or any other clinically significant illness within two weeks of dose administration
* History of gastrointestinal disease including inflammatory bowel disease, peptic ulcer disease, gastrointestinal hemorrhage
* Inadequate hematologic, renal or liver function
* Positive for hepatitis A, hepatitis B, hepatitis C, or HIV infection
* History (within 3 months of screening) of alcohol consumption exceeding 14 units per week on average (1 unit = 10 grams of alcohol). Alcohol consumption will be prohibited at least 48 hours before screening, 48 hours before admission, 48 hours after each dose, and 48 hours before each scheduled visit
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Subjects who had received IFN or peginterferon within 8 weeks prior to dosing
* Participation in other clinical studies of a new chemical entity within 60 days prior to study randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to 44 days

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose and up to 48 hours post-dose
Pharmacokinetics: Maximum plasma concentration (Cmax) | Pre-dose and up to 48 hours post-dose
Effect of food on pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose and up to 48 hours post-dose
Pharmacodynamics: Cytokines/neopterin levels | Pre-dose and up to 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands